CLINICAL TRIAL: NCT03294018
Title: Heart Rate Changes Following the Administration of Sugammadex
Status: Completed | Type: Observational
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chairman, Professor of Anesthesiology, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB17-00540
Record Dates: First submitted 2017-09-22; First posted 2017-09-26 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bradycardia during sugammadex administration: Recording any heart rate changes during planned administration of sugammadex.
  Interventions: Other: Recording heart rate changes

INTERVENTIONS:
Other: Recording heart rate changes — Recording heart rate changes during planned sugammadex administration.

SUMMARY:
This a prospective study when the clinician decides to use sugammadex, heart rate will be recorded every minute for 15 minutes following its administration. If bradycardia occurs and a clinical decision is made to treat it, the medications and doses used will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 0-18 years
* Anesthetic plan includes NMB reversal with sugammadex

Exclusion Criteria:

* Sugammadex not used during the case

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male and female 0-18 years old undergoing surgery with anesthetic plan with sugammadex.
Sampling Method: Non-Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Bradycardia during sugammadex administration | intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States